CLINICAL TRIAL: NCT00420420
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial to Evaluate the Safety and Efficacy of MK0249 for the Symptomatic Treatment of Alzheimer's Disease
Brief Title: MK0249 for the Symptomatic Treatment of Alzheimer's Disease (MK0249-011)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0249-011; 2006_534
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — MK-0249

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MK0249 (Experimental)
  Interventions: Drug: MK0249
- placebo (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: MK0249 — MK0249 two (2) 2.5 mg capsules quaque die (qd) for 28 day treatment period.
  Arms: MK0249
Drug: Comparator: Placebo (unspecified) — MK0249 two (2) 2.5 mg Pbo capsules qd for a 28 day treatment period
  Arms: placebo

SUMMARY:
The purpose of this study is to test the efficacy and safety of an investigational medication for improving symptoms of Alzheimer's Disease. Subjects will receive either active medication or placebo for 28 days. Tests of memory, concentration will be included. Safety will be monitored using routine clinical and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or females
* Age at least 55 years or older
* Mild-to-moderate Alzheimer's Disease, with Mini Mental State Examination (MMSE) between 18 and 26, inclusive, Modified Hachinski Ischemic Scale (MHIS) score =/<4, Global CDR score of 1 or 2, and who have a reliable informant/caregiver to accompany patient to all clinic visits
* If using symptomatic Alzheimer's Disease treatments, patients must be on the medication for 3 months and on a STABLE DOSE for at least 2 months

Exclusion Criteria:

* Patients cannot be living in a skilled nursing facility
* Patients cannot have poorly-controlled hypertension
* Patients cannot have the following conditions within 6 months of screening: significant cardiovascular disorders, active major depressive disorder, gastroesophageal reflux disease (GERD), or clinically significant sleep disorder
* Various concomitant therapy restrictions

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Egan M, Yaari R, Liu L, Ryan M, Peng Y, Lines C, Michelson D. Pilot randomized controlled study of a histamine receptor inverse agonist in the symptomatic treatment of AD. Curr Alzheimer Res. 2012 May;9(4):481-90. doi: 10.2174/156720512800492530. PMID 22272611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Dosed: 13 JAN 2007; Last Patient Last Treatment: 14 AUG 2008. 15 U.S. outpatient centers.
Pre-assignment Details: At Visit 1, patients were assessed using the protocol inclusion and exclusion criteria, then, if deemed eligible, patients were randomized at Visit 3.
Groups:
- MK0249 (5 mg): Patients were randomly assigned to 28 days of treatment with 5 mg MK-0249 taken orally daily (qd).
- Placebo: Patients were randomly assigned to 28 days of treatment with matching placebo taken orally daily (qd).
Period: Overall Study
Arm/Group | MK0249 (5 mg) | Placebo
Started | 73 (Number of patients randomized.) | 71 (Number of patients randomized.)
Completed | 65 (One patient from the MK-0249 arm discontinued the trial due to an AE prior to receiving study drug.) | 67
Not Completed | 8 | 4
Not completed — Adverse Event | 5 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — sponsor decision (abnormal ECG @ screen) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0249 (5 mg) | Placebo | Total
Number analyzed (Participants) | 73 | 71 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (6.91) | 73.7 (8.91) | 74.05 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 36 | 79
  Male | 30 | 35 | 65

OUTCOME MEASURES:

1. Primary Outcome: Week 4 Change From Baseline in Computerized Neuropsychological Test Battery (CNTB): Short CNTB Summary Score.
Description: The CNTB was used to evaluate cognitive function, as measured by the mean change from Baseline to Week 4 in the short CNTB summary score. The short CNTB summary score was scored as the mean score across 5 modules: Word List Learning-Selective Reminding, Word List Learning-Delayed Recall, Simple Reaction Time, Choice Reaction Time, and Visual Memory subtests. The short CNTB summary score ranges from 0 to 100, with higher scores (and positive changes from baseline) indicating better performance.
Time Frame: Baseline and Week 4
Population: Full Analysis Set: All patients who were randomized, took at least one dose of study medication, and had at least one efficacy measurement at either Baseline, Week 2 or Week 4. Patients were counted in the treatment group to which they were randomized.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MK0249 (5 mg) | Placebo
Number analyzed (Participants) | 59 | 62
units on a scale | 0.13 (0.61) | -0.76 (0.57)
Statistical Analysis 1: Comparison: MK0249 (5 mg) vs Placebo; comparison at Week 4; Test type: Superiority or Other; p = 0.283, Mixed Models Analysis — A longitudinal mixed model was used to compare groups, including factors for week, strata (MMSE score and concomitant AD therapy), treatment, and week-by-treatment interaction

2. Secondary Outcome: Week 4 Change From Baseline in Cognition Summary Score (CSS)
Description: The CSS was used to evaluate cognitive function as measured by the mean change from Baseline to Week 4 in the CSS total score. The CSS was derived from the correct sequence percentage from the Route Test and 6 of the CNTB scores (the CSS was scored as the mean of the 7 scores). CSS scores can range from 0 to 100, higher scores (and positive changes from baseline) indicate better performance.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MK0249 (5 mg) | Placebo
Number analyzed (Participants) | 49 | 51
units on a scale | 1.19 (0.75) | -0.19 (0.72)
Statistical Analysis 1: Comparison: MK0249 (5 mg) vs Placebo; comparison at week 4; Test type: Superiority or Other; p = 0.180, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Week 4 Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog): ADAS-Cog Total Score
Description: The ADAS-Cog, scored as the total score of 11 tasks including mazes was used to evaluate cognitive function, as measured by the mean change from Baseline to Week 4 in the ADAS-Cog total score. The ADAS-Cog total score ranges from 0 to 70, with higher total scores indicating more impairment. Lower scores (and negative changes from Baseline) indicate better performance.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MK0249 (5 mg) | Placebo
Number analyzed (Participants) | 70 | 68
units on a scale | -1.42 (0.50) | -1.17 (0.49)
Statistical Analysis 1: Comparison: MK0249 (5 mg) vs Placebo; comparison at Week 4; Test type: Superiority or Other; p = 0.716, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Baseline: Short CNTB Summary Score.
Description: as for outcome 1
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MK0249 (5 mg) | Placebo
Number analyzed (Participants) | 64 | 68
units on a scale | 35.98 (5.72) | 36.23 (6.59)

5. Other Pre Specified Outcome: Baseline: ADAS-Cog Total Score
Description: as for outcome 3
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MK0249 (5 mg) | Placebo
Number analyzed (Participants) | 73 | 70
units on a scale | 19.08 (7.51) | 18.42 (7.32)

6. Other Pre Specified Outcome: Baseline: Cognition Summary Score (CSS)
Description: as for outcome 2
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MK0249 (5 mg) | Placebo
Number analyzed (Participants) | 56 | 57
units on a scale | 42.31 (7.35) | 43.79 (7.32)

ADVERSE EVENTS:
Time Frame: Patients were assessed for AEs from Visit 2 (Day 0) Baseline through Visit 8 (Day 43) Post-Study Safety Visit.
Arm/Group | MK0249 (5 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 3/73 | 1/70
Other Adverse Events (participants affected / at risk) | 29/73 | 9/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0249 (5 mg) (N=73) | Placebo (N=70)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK0249 (5 mg) (N=73) | Placebo (N=70)
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Stomach discomfort (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 3
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 6 | 1
Insomnia (Psychiatric disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.